CLINICAL TRIAL: NCT05394688
Title: Directional Deep Brain Stimulation in Advanced Parkinson's Disease - Clinical Review
Brief Title: Directional Deep Brain Stimulation With Patients With Advanced Parkinson's Disease
Acronym: dDBS
Status: Completed | Type: Observational
Sponsor: Hospital District of Helsinki and Uusimaa (Other)
Responsible Party: Principal Investigator, Maija Koivu, M.D., Specialist in Neurology, Hospital District of Helsinki and Uusimaa
Other Study IDs: HospitalIDHU
Record Dates: First submitted 2020-09-28; First posted 2022-05-27 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease
Keywords: deep brain stimulation; advanced Parkinson's disease; DBS; dDBS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess the clinical outcome in patients with Parkinson's disease treated with directional deep brain stimulation (dDBS). The patients have been selected for the dDBS treatment by their treating neurologist. The study is a registry-based follow-up study.

DETAILED DESCRIPTION:
The study group consists of patients with advanced Parkinson's disease treated with directional deep brain stimulation in Helsinki University Hospital between 2017 - 2020. The study is a registry-based follow-up study. The aim of the study is to assess the clinical outcome and possible adverse effects of the dDBS treatment. The data will be collected from the patient records. The observed time points are 6-month's, 12-month's and 18-month's postoperative visits.

The following data will collected: the scores of Unified Parkinson's disease questionnaire part III (UPDRS-III), Non-Motor Symptoms Questionnaire (NMS-quest), Beck Depression Inventory (BDI), Mini-Mental State Examination (MMSE), Abnormal Involuntary Movement Scale (AIMS) evaluated in the screening phase for dDBS treatment and at 6-months' follow-up. Possible levodopa equivalent dose changes, LEDDs, will also be assessed at these time points.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced Parkinson's disease and treated with directional deep brain stimulation

Exclusion Criteria:

* patients with advanced Parkinson's disease and not treated with directional deeb brain stimulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of the initial 63 patients with Parkinson'd disease treated with directional deep brain stimulation in Helsinki University Hospital
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The actual use of directional DBS stimulation in everyday life during the follow-up | 6-18 months
  The use of directionality in DBS in patients with PD in everyday life

SECONDARY OUTCOMES:
The changes of UPDRS part III score during the DBS treatment | From the initiation of DBS treatment to 18-month's postoperative visit
  The changes of UPDRS part III score during the DBS treatment
Evaluation of the dDBS parameters | 6 months to 18 months
  The use of dDBS, active contacts and the dDBS programming protocol will be studied.
Possible adverse effects | 6 months-18 months
  Possible adverse effects of dDBS operation and treatment will be collected
LEDDs | From preoperative visit to 18 month's postoperative visit
  Possible changes of levodopa equivalent doses, LEDDs, are studied

CONTACTS AND LOCATIONS:
Overall Officials: Eero Pekkonen, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- HUH Meilahti Hospital, department of neurology, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weaver FM, Follett K, Stern M, Hur K, Harris C, Marks WJ Jr, Rothlind J, Sagher O, Reda D, Moy CS, Pahwa R, Burchiel K, Hogarth P, Lai EC, Duda JE, Holloway K, Samii A, Horn S, Bronstein J, Stoner G, Heemskerk J, Huang GD; CSP 468 Study Group. Bilateral deep brain stimulation vs best medical therapy for patients with advanced Parkinson disease: a randomized controlled trial. JAMA. 2009 Jan 7;301(1):63-73. doi: 10.1001/jama.2008.929. PMID 19126811
- [Background] Deuschl G, Schade-Brittinger C, Krack P, Volkmann J, Schafer H, Botzel K, Daniels C, Deutschlander A, Dillmann U, Eisner W, Gruber D, Hamel W, Herzog J, Hilker R, Klebe S, Kloss M, Koy J, Krause M, Kupsch A, Lorenz D, Lorenzl S, Mehdorn HM, Moringlane JR, Oertel W, Pinsker MO, Reichmann H, Reuss A, Schneider GH, Schnitzler A, Steude U, Sturm V, Timmermann L, Tronnier V, Trottenberg T, Wojtecki L, Wolf E, Poewe W, Voges J; German Parkinson Study Group, Neurostimulation Section. A randomized trial of deep-brain stimulation for Parkinson's disease. N Engl J Med. 2006 Aug 31;355(9):896-908. doi: 10.1056/NEJMoa060281. PMID 16943402
- [Result] Steigerwald F, Muller L, Johannes S, Matthies C, Volkmann J. Directional deep brain stimulation of the subthalamic nucleus: A pilot study using a novel neurostimulation device. Mov Disord. 2016 Aug;31(8):1240-3. doi: 10.1002/mds.26669. Epub 2016 May 31. PMID 27241197
- [Result] Dembek TA, Reker P, Visser-Vandewalle V, Wirths J, Treuer H, Klehr M, Roediger J, Dafsari HS, Barbe MT, Timmermann L. Directional DBS increases side-effect thresholds-A prospective, double-blind trial. Mov Disord. 2017 Oct;32(10):1380-1388. doi: 10.1002/mds.27093. Epub 2017 Aug 26. PMID 28843009
- [Result] Contarino MF, Bour LJ, Verhagen R, Lourens MA, de Bie RM, van den Munckhof P, Schuurman PR. Directional steering: A novel approach to deep brain stimulation. Neurology. 2014 Sep 23;83(13):1163-9. doi: 10.1212/WNL.0000000000000823. Epub 2014 Aug 22. PMID 25150285
- [Result] Schnitzler A, Mir P, Brodsky MA, Verhagen L, Groppa S, Alvarez R, Evans A, Blazquez M, Nagel S, Pilitsis JG, Potter-Nerger M, Tse W, Almeida L, Tomycz N, Jimenez-Shahed J, Libionka W, Carrillo F, Hartmann CJ, Groiss SJ, Glaser M, Defresne F, Karst E, Cheeran B, Vesper J; PROGRESS Study Investigators. Directional Deep Brain Stimulation for Parkinson's Disease: Results of an International Crossover Study With Randomized, Double-Blind Primary Endpoint. Neuromodulation. 2022 Aug;25(6):817-828. doi: 10.1111/ner.13407. Epub 2022 Feb 2. PMID 34047410
- [Result] Rammo RA, Ozinga SJ, White A, Nagel SJ, Machado AG, Pallavaram S, Cheeran BJ, Walter BL. Directional Stimulation in Parkinson's Disease and Essential Tremor: The Cleveland Clinic Experience. Neuromodulation. 2022 Aug;25(6):829-835. doi: 10.1111/ner.13374. Epub 2022 Jun 14. PMID 33733515